CLINICAL TRIAL: NCT05510843
Title: An Open-label, Multicenter Study to Assess the Safety, Pharmacokinetics and Pharmacodynamic Effects of THB001 in Adult Patients With Chronic Cold Urticaria
Brief Title: A Study to Evaluate THB001 in Adult Patients With Chronic Cold Urticaria
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision to discontinue the study was made after observing moderate drug induced liver injury in two subjects enrolled in the first dose cohort.
Sponsor: Third Harmonic Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: THB001-01-002
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Chronic Cold Urticaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- THB001 Dose Level A (Experimental)
  Interventions: Drug: THB001
- THB001 Dose Level B (Experimental)
  Interventions: Drug: THB001
- THB001 Dose Level C (Experimental)
  Interventions: Drug: THB001

INTERVENTIONS:
Drug: THB001 — 100 mg capsules for oral administration

SUMMARY:
This is a phase 1b, open label, non-randomized, sequential dose-escalation, multicenter trial in adult patients with chronic cold urticaria.

ELIGIBILITY:
Key Inclusion Criteria:

1. Women and Men ages 18-75
2. Diagnosed with chronic, cold inducible urticaria for at least 3 months prior to starting the study and refractory to antihistamine treatment
3. Positive cold stimulation test assessed by TempTest® at the Screening and Baseline visits
4. Considered healthy as assessed by medical evaluation including review of medical history, physical examination, vital signs, laboratory tests and ECG recording
5. Willing and able to participate in all visits, undergo all study procedures and adhere to study restrictions

Key Exclusion Criteria:

1. A diagnosis of acute urticaria or non-cold chronic inducible urticaria
2. Ongoing treatment with immunosuppressant drugs (corticosteroids, cyclosporine, azathioprine, methotrexate, omalizumab, dupilumab, sulfasala-zine, dapsone or others)
3. A positive test for pregnancy, HIV, Hepatitis B or Hepatitis C
4. Clinical laboratory values outside of the normal ranges at the Screening visit
5. History of any clinically significant abnormality that would contraindicate participation

There are additional criteria that your study doctor will review with you to confirm you are eligible for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by the incidence and severity of adverse events | From Day 1 through Week 12
  Safety evaluations will include analyses of adverse events by treatment group

CONTACTS AND LOCATIONS:
Locations (2):
- Charité - Universitätsmedizin Berlin Institute of Allergology, Berlin, Germany
- Centre for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Results of safety (AEs, SAEs) will be made available.
Time Frame: Within 1 year after last subject last visit.